CLINICAL TRIAL: NCT00752791
Title: A Phase 2 Study of the Safety and Efficacy of Hematide Injection for the Maintenance Treatment of Anemia in Peritoneal Dialysis Subjects Previously Treated With Epoetin
Brief Title: Efficacy and Safety of Peginesatide Injection for the Maintenance Treatment of Anemia in Peritoneal Dialysis Participants Previously Treated With Epoetin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX01_201; 2008-003458-13 (EudraCT Number); U1111-1114-0301 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Anemia
Keywords: Anemia; Drug Therapy; Peritoneal Dialysis.
MeSH Terms: conditions — Anemia | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginesatide (Experimental)
  Interventions: Drug: Peginesatide

INTERVENTIONS:
Drug: Peginesatide — Peginesatide 0.04 to 0.16 mg/kg, subcutaneous injection, once every 4 weeks for up to 25 weeks. Initial dose based on patient's previous total weekly Epoetin dose, and thereafter could be adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline.
  Other Names: Hematide; AF37702; Omontys

SUMMARY:
The purpose of this study is to determine the efficacy and safety of peginesatide injection for maintenance treatment of anemia in participants on peritoneal dialysis.

DETAILED DESCRIPTION:
According to the International Federation of Renal Registries, in 1999 the prevalence of peritoneal dialysis in the United States as approximately 9.5% of patients receiving dialysis (2005 United States Renal Data Systems data indicates a prevalence of around 7.5%). Data from Europe in 1999 to 2000 (not including the United Kingdom, France or Germany) indicated peritoneal dialysis was the mode of dialysis in approximately 11.1% of dialysis patients. 2006 data from the United Kingdom indicates that more than 20% of patients on dialysis are receiving peritoneal dialysis while French and German data indicate rates of 8.1% and 4.8% respectively. More than 90% of patients with chronic renal failure/chronic kidney disease Stage 5 (End Stage Renal Disease) are anemic. The vast majority of patients receiving hemodialysis or peritoneal dialysis receive erythropoiesis-stimulating agent therapy to treat their anemia.

Anemia of chronic renal failure is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors also include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The prevalence of anemia increases with progressive deterioration of renal function, and affects more than 90% of patients with chronic kidney disease (CKD) Stage 5 (End Stage Renal Disease). Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function and exercise capacity, increased left ventricular hypertrophy and heart failure. Treatment of anemia reduces morbidity and mortality risks and may improve quality of life.

Erythropoiesis stimulating agents have been established as a treatment for anemia in chronic renal failure participants, and have improved the management of anemia over alternatives such as transfusion. Peginesatide (hematide) is a parenteral formulation being developed for the correction of anemia in patients with chronic renal failure, and binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Participants in this study received variable doses of peginesatide injection once every four weeks. Total commitment time for this study was about 29 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was a man or woman and 18 to 90 years of age, inclusive.
2. The patient had CKD and had been on peritoneal dialysis for ≥3 months before enrollment.
3. The patient was on stable SC epoetin (alfa or beta) maintenance therapy continuously prescribed for a minimum of 8 weeks prior to enrollment.
4. The patient had 4 consecutive Hb values with a mean ≥10.0 and ≤12.0 g/dL during the screening period, with the difference between the mean of the first confirmed (2 consecutive) Hb values and the mean of the last confirmed (2 consecutive) Hb values being ≤1.0 g/dL.
5. The patient had 1 ferritin level ≥100 ng/mL within 4 weeks before enrollment.

Exclusion Criteria:

1. The patient had known bleeding or coagulation disorder.
2. The patient had known hematologic disease or cause of anemia other than renal disease (e.g., pure red cell aplasia, homozygous sickle-cell disease, thalassemia, multiple myeloma, hemolytic anemia, and myelodysplastic syndrome).
3. The patient had received a recent course of intensive iron replacement (i.e., more than 500 mg IV in the 28 days before enrollment).
4. The patient had advanced chronic congestive heart failure defined by New York Heart Association Class III or IV.
5. The patient had a known history of seizure disorder or received antiepileptic medication for a seizure disorder within 6 months before enrollment.
6. The patient had a scheduled kidney transplant. (Note: patients who were currently on a transplant waiting list were not excluded unless there was an identified donor).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (23):
- United States (19):
  - Azusa, California
  - Los Angeles, California
  - Whittier, California
  - Naples, Florida
  - Decatur, Georgia
  - Evergreen Park, Illinois
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - New Iberia, Louisiana
  - Shreveport, Louisiana
  - Columbus, Mississippi
  - Tupelo, Mississippi
  - New York, New York
  - Williamsville, New York
  - Canton, Ohio
  - Arlington, Texas
  - Tyler, Texas
  - Fairfax, Virginia
  - Mechanicsville, Virginia
- New Lambtom, New South Wales, Australia
- Modena, Modena, Italy
- Dunedin, Dunedin, New Zealand
- London, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 26 sites in Australia, Italy, New Zealand, the United Kingdom and the United States from 31 October 2008 to 19 May 2010.
Pre-assignment Details: Participants with chronic renal failure on peritoneal dialysis and receiving stable Epoetin (alfa or beta) maintenance therapy were enrolled into 1 treatment group (peginesatide injection).
Period: Overall Study
Arm/Group | Peginesatide
Started | 59
Completed | 43
Not Completed | 16
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Death | 1
Not completed — Renal transplant | 3
Not completed — Switched to hemodialysis | 2
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (15.99)
Age, Customized [Number; unit: participants]
  <65 years | 42
  ≥65 to <75 years | 10
  ≥75 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The primary efficacy endpoint was the mean change in Hemoglobin between Baseline (the mean of the 4 most recent hemoglobin values prior to Enrollment and the hemoglobin on the day of Enrollment) and the Evaluation Period (mean hemoglobin from Weeks 20 to 25).
Time Frame: Baseline and Week 20 to Week 25.
Population: The Full Analysis Set included all patients who received at least 1 dose of peginesatide injection and where data was available at both time points (indicated by N).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
g/dL
  Baseline [N=59] | 11.22 (0.495)
  Evaluation Period [N=46] | 11.33 (1.066)
  Change from Baseline [N=46] | 0.10 (1.154)
Statistical Analysis 1: Comparison: Peginesatide; Test type: Superiority or Other; Mean change from Baseline = 0.10, 95% CI 2-sided [-0.24 to 0.44] — A two-sided 95% CI of the estimated mean change from Baseline in hemoglobin was derived from the t-distribution

2. Secondary Outcome: Percentage of Participants With Hemoglobin Within the Target Range of 10.0 to 12.0 g/dL During the Evaluation Period
Description: Mean hemoglobin was calculated from measurements taken during the Evaluation Period (Week 20 to Week 25). The target hemoglobin range was 10.0 to 12.0 g/dL.
  The 95% confidence interval was calculated from the normal approximation with continuity correction.
Time Frame: Week 20 to Week 25.
Population: Full analysis set where data was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 46
percentage of participants | 63.0 [48.0 to 78.1]

3. Secondary Outcome: Percentage of Participants With a Change in Hemoglobin From Baseline to the Evaluation Period Within 1 g/dL
Description: Percentage of participants with a mean change in Hemoglobin between Baseline (the mean of the 4 most recent hemoglobin values prior to enrollment and the hemoglobin on the day of enrollment) and the Evaluation Period (mean hemoglobin from measured at Weeks 20 to 25) of less than or equal ± 1 g/dL. The 95% confidence interval was calculated from the normal approximation with continuity correction.
Time Frame: Baseline and Week 20 to Week 25.
Population: Full analysis set where data was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 46
percentage of participants | 60.9 [45.7 to 76.1]

4. Secondary Outcome: Percentage of Participants With Red Blood Cell Transfusions
Description: The percentage of participants who received one or more red blood cell transfusions, including packed red blood cells and whole blood transfusions, during the Titration Period (Weeks 1 - 19) and Evaluation Period (Weeks 20 -25). 95% Confidence Intervals were calculated from the normal approximation with continuity correction. One patient had the last study visit during the titration period and the transfusion after the titration period. This patient is excluded from the summary of evaluation period.
Time Frame: Up to 25 weeks.
Population: Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
percentage of participants
  Entire study (n=59) | 10.2 [1.6 to 18.7]
  Titration Period (n=59) | 5.1 [0.0 to 11.5]
  Evaluation period (n=47) | 4.3 [0.0 to 11.1]

5. Secondary Outcome: Mean Hemoglobin During 4-week Intervals
Description: Hemoglobin was measured every 2 weeks during the Titration Period (Weeks 1-19) and weekly during the Evaluation Period (Weeks 20-25). One patient did not have central lab hemoglobin value during a regularly scheduled visit during weeks 2-5.
Time Frame: Up to 25 weeks.
Population: Full Analysis Set where data was available for each time interval (indicated by N).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
g/dL
  Week 2-5 [N=58] | 11.57 (0.741)
  Week 6-9 [N=56] | 11.65 (1.044)
  Week 10-13 [N=54] | 11.53 (1.119)
  Week 14-17 [N=52] | 11.33 (1.037)
  Week 18-21 [N=45] | 11.46 (1.004)
  Week 22-25 [N=46] | 11.25 (1.122)

6. Secondary Outcome: Percentage of Participants With Target Hemoglobin of 10.0 to 12.0 g/dL by 4-week Intervals
Description: Percentage of participants with mean hemoglobin levels falling between the target level of 10.0 to 12.0 g/dL during 4-week study intervals. Hemoglobin was measured every 2 weeks during the Titration Period (Weeks 1-19) and weekly during the Evaluation Period (Weeks 20-25). 95% Confidence Intervals were calculated from the normal approximation with continuity correction.
Time Frame: Up to 25 weeks.
Population: Full analysis set where data was available for each time interval (indicated by N).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
percentage of participants
  Week 2-5 [N=58] | 67.2 [54.3 to 80.2]
  Week 6-9 [N=56] | 53.6 [39.6 to 67.5]
  Week 10-13 [N=54] | 59.3 [45.2 to 73.3]
  Week 14-17 [N=52] | 61.5 [47.4 to 75.7]
  Week 18-21 [N=45] | 64.4 [49.3 to 79.5]
  Week 22-25 [N=46] | 63.0 [48.0 to 78.1]

7. Secondary Outcome: Percentage of Participants With Dose Adjustments During the Study
Description: The peginesatide dose was adjusted to maintain hemoglobin values in the target range of 10 to 12 g/dL and ±1.5 g/dL from Baseline during the Titration Period (Weeks 1-19) and Evaluation Period (Weeks 20-25). A dose was classified as adjusted if it was not within 20% of the previous dose. A dose was classified as increased or decreased if it was >20% higher or >20% lower respectively, than the previous dose.
Time Frame: From Week 4 to Week 25
Population: Safety Analysis Set. N indicates the number of patients with study drug administered during the period after excluding the initial dose of study drug and excluding the first dose after a restart of study drug and is the denominator for percentage calculations.
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 59
percentage of participants
  Any adjustment in Titration Period [N=57] | 80.7
  Any adjustment in Evaluation Period [N=42] | 52.4
  Dose increased in Titration Period [N=57] | 28.1
  Dose increased in Evaluation Period [N=42] | 16.7
  Dose decreased in Titration Period [N=57] | 66.7
  Dose decreased in Evaluation Period [N=42] | 35.7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that occurred on or after the day of the first dose of peginesatide injection through the Follow-up phone call, which occurred within 28 days after the last dose.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Peginesatide
Serious Adverse Events (participants affected / at risk) | 27/59
Other Adverse Events (participants affected / at risk) | 41/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=59)
Leukocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1 — This treatment emergent death occurred during titration period and is considered related.
Ventricular fibrillation (Cardiac disorders) | 1
Peritonitis (Gastrointestinal disorders) | 9 — This treatment-emergent death occured during titration period and is not related.
Colonic polyp (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Medical device complication (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Fungal peritonitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1 — This treatment-emergent death occured during evaluation period period and is not related.
Septic shock (Infections and infestations) | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1 — This treatment-emergent death was reported 74 days after last dose of study drug and is considered related to study drug.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pseudoporphyria (Skin and subcutaneous tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=59)
Diarrhoea (Gastrointestinal disorders) | 9
Peritonitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Oedema Peripheral (General disorders) | 5
Urinary Tract Infection (Infections and infestations) | 5
Catheter Site Infection (Infections and infestations) | 4
Nasopharygitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 3
Excoriation (Injury, poisoning and procedural complications) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.